CLINICAL TRIAL: NCT04584021
Title: Pilot Project Based on the Use of Wearable Devices to Assess the Impact of Stress in the Work Environment on the Quality of Life of Workers: Project SQoF-WEAR
Brief Title: Use of Wearable Devices to Assess the Impact of Stress in Workers' Life Quality
Acronym: SQoF-WEAR
Status: Completed | Type: Observational
Sponsor: Universidade da Coruña (Other)
Collaborators: Center on Information and Communication Technologies (Other); Universidade do Porto (Other)
Responsible Party: Principal Investigator, Javier Pereira, Professor PhD, Universidade da Coruña
Other Study IDs: 2019/249
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Stress Disorder; Burnout, Professional; Sleep Disorder; Quality of Life; Anxiety State
Keywords: Stress Disorder; Burnout; Participatory Health; Quality of life; Daily functioning
MeSH Terms: conditions — Stress Disorders, Traumatic; Burnout, Professional; Sleep Wake Disorders; Anxiety Disorders; Burnout, Psychological

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stress study participants: Adults who reported stress problems derived from work
  Interventions: Device: Xiaomi MiBand3; Other: Socio-demographic questionnaire; Other: EuroQol-5D-5L; Other: Pittsburgh Sleep Quality Index (PSQI); Other: State-Trait Anxiety Inventory (STAI); Other: Perceived Stress Scale-10 (PSS-10); Other: Stress questionnaire

INTERVENTIONS:
Device: Xiaomi MiBand3 — Recording of sleep, activity and heart rate data to study their association with stress.
Other: Socio-demographic questionnaire — Self-made questionnaire to be filled by the participants at the beginning of the study with the following personal data: age, gender, marital status, residential environment, cohabitation unit, educational level, socio-economic level, contract, working hours, overtime or not, number of overtime hours in a day, overtime frequency and perceived stress level
Other: EuroQol-5D-5L — Quality of life questionnaire to be filled by the participants at the beginning, mid-term and completion of the study with the following information: severity index, social value index for each health condition. Subjective evaluation of health status from 0 to 100.
Other: Pittsburgh Sleep Quality Index (PSQI) — Questionnaire to be filled by the participants whose outcome is the perceived quality, quantity and efficient of sleep. To be given at the beginning, mid-term, and completion of the study.
Other: State-Trait Anxiety Inventory (STAI) — Questionnaire to be filled by the participants which measures the anxiety level. To be given at the beginning, mid-term and completion of the study.
Other: Perceived Stress Scale-10 (PSS-10) — Questionnaire to be filled by the participants which measures the stress level. To be given at the beginning, mid-term and completion of the study.
Other: Stress questionnaire — Questionnaire designed by a work stress psychologist professional from the research group which is focused on stress and daily functioning. This questionnaire was given for the participants to fill. It is composed by 3 daily items and 4 weekly items.

SUMMARY:
Introduction: Work stress has become more and more important in the last years as it affects both health and productivity of workers. In the last years, different wearables devices have started to be used to monitor stress at work to understand their consequences on daily life activity and sleep quality.

Objective: to establish whether wearable wristbands are devices capable of determining the work stress level of workers from a research center in Galicia, for which different variables related to the work stress level and quality of life of these workers will be evaluated.

Methods and analysis: The only inclusion criterion is to be a worker from a research center from Galicia. As for exclusion criteria, will not be allowed to participate those workers who are close to retirement ( <5 years), have health issues that hinder participation in the study, or present skin hypersensitivity or allergic reactions due to the materials the wristbands are made.

This is a pilot study to determine the viability, sample size, cost, and duration of the study. This is an observational, analytic, and longitudinal study. In other words, in this study different variables from the population of interest will be observed and recorded without any direct intervention, so as to establish causality associations between these variables. It is considered as longitudinal since a six-months tracking of the variables will be performed.

As for the statistical analysis, different tests will be performed to analyse the distribution, correlation, and association of the different features, as well as the significant differences between them at different points of the study (detailed below).

DETAILED DESCRIPTION:
Introduction: Stress is a natural phenomenon within the human body that prepares the organism for action. However, due to the current life and work habits and demands, stress goes beyond what is beneficial and starts to suppose a burden. Nowadays, work stress, which is defined as "a harmful reaction, which people have to deal with, to the pressures and undue demands placed on them at work", has gained importance as it affects both health and productivity of workers. If stress persists over time, it can lead to the syndrome known as Burnout, which implies deep exhaustion, and inefficiency. In the last years, different wearable devices have started to be used to monitor stress at work with the aim of understanding their consequences on physical activity and sleep quality.

Objective: To establish whether wearable wristbands are devices capable of determining the work stress level of workers from a research center in Galicia. To this end, it will be determined the work stress level and quality of life of these workers to conclude if the devices measure the work stress with precision. Also, different physical activity, sleep and occupational functioning patterns will be identified to study the relation between them and the work stress level and quality of life.

Methods and Analysis: The study will be carried out with workers from a research center from Galicia, being this the only inclusion criterion. As for exclusion criteria, workers will not be allowed to participate if they are expected to retire in a period of 5 years or less, have significant health issues that hinder the participation in the study, or present skin hypersensitivity or allergic reactions caused by the materials the wristbands are made of.

This is a pilot study to determine the viability, sample size, cost, and duration of the study. Likewise, a pilot project has also been designed in this study in order to "demonstrate that the planned measurements, the data collection instruments and the data management system are feasible and effective". This is an observational, analytical, and longitudinal study. That is, in this study different variables of the population under study will be observed and recorded without intervention and with the aim of establishing causal associations between variables. It is considered longitudinal because variables will be followed for 6 months, continuously recording and monitoring physical activity and the quality of sleep (wristbands), and in a specific way, variables related to work stress, quality of life, and perception of the quality of sleep and the level of physical activity (specific evaluation tools).

As for the statistical analysis, and once the data are preprocessed, for the collected variables the Kolmogorov-Smirnov will be applied to check if they behave as a normal distribution. Otherwise, posterior analysis with non-parametric tests will be performed. The correlation of the numeric variables will be analysed through the Pearson or Spearman's Rho correlation depending on the sample distribution. A Chi-Square test will be used to assess the association between categoric variables unless the observed frequencies are <5%, for which a likelihood ratio test would be used. Regarding the association between quantitative and qualitative variables, the mean comparison with a T and ANOVA test, or a Mann Whitney and Kruskal Wallis test, as appropriate, will be performed. To finish, with the aim of determining whether there are significant differences between the results of the beginning, mid-term and final evaluations, a Wilcoxon test will be applied.

ELIGIBILITY:
Inclusion Criteria:

* To be developing their professional activity in a research center

Exclusion Criteria:

* To be close to retirement (5 years or less)
* To have significant health condition complications that difficult active participation in the study
* To present hypersensitivity in the skin or a recognized allergy to the material of which are made the cases or straps of the wearable wristbands to be used as one of the measuring instruments of the study are made.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Working population in a research center, who accept and consent to participate in a stress project.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Stress and anxiety level | Until the completion of the study (around 12 months)
  Influence of stress and anxiety in the worker

SECONDARY OUTCOMES:
Sleep recording | Until the completion of the study (around 12 months)
  Measured by the Xiaomi MiBand3
Physical activity tracking | Until the completion of the study (around 12 months)
  Measured by the Xiaomi MiBand3
Quality of life self-perception | At the beginning, mid-term and completion of the study
  Measured by the EuroQol-5D-5L scale
Sleep habits | At the beginning, mid-term and completion of the study
  Measured by the Pittsburgh Sleep Quality Index (PSQI)
Anxiety self-perception | At the beginning, mid-term and completion of the study
  Measured by the State-Trait Anxiety Inventory (STAI)
Stress self-perception | At the beginning, mid-term and completion of the study
  Measured by the Perceived Stress Scale-10 (PSS-10)
Stress influence on daily functioning | Until the completion of the study (around 12 months)
  Measured by the stress questionnaire designed by a work stress psychologist professional

CONTACTS AND LOCATIONS:
Overall Officials: Javier Pereira, PhD, Principal Investigator — Universidade da Coruña
Locations (1):
- Universidade da Coruña, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Almeida DM. Resilience and vulnerability to daily stressors assessed via diary methods. Curr Dir Psychol Sci. 2005 Apr 1;14(2):64-8
- [Background] Almeida DM, Wethington E, Kessler RC. The daily inventory of stressful events: an interview-based approach for measuring daily stressors. Assessment. 2002 Mar;9(1):41-55. doi: 10.1177/1073191102091006. PMID 11911234
- [Background] Bhui K, Dinos S, Galant-Miecznikowska M, de Jongh B, Stansfeld S. Perceptions of work stress causes and effective interventions in employees working in public, private and non-governmental organisations: a qualitative study. BJPsych Bull. 2016 Dec;40(6):318-325. doi: 10.1192/pb.bp.115.050823. PMID 28377811
- [Background] Maslach C, Schaufeli WB, Leiter MP. Job burnout. Annu Rev Psychol. 2001;52:397-422. doi: 10.1146/annurev.psych.52.1.397. PMID 11148311
- [Background] Estevez-Mujica CP, Quintane E. E-mail communication patterns and job burnout. PLoS One. 2018 Mar 8;13(3):e0193966. doi: 10.1371/journal.pone.0193966. eCollection 2018. PMID 29518128
- [Background] Hogan V, Hogan M, Hodgins M. A study of workaholism in Irish academics. Occup Med (Lond). 2016 Aug;66(6):460-5. doi: 10.1093/occmed/kqw032. Epub 2016 May 11. PMID 27170737
- [Background] Pignata S, Winefield AH. Stress-reduction interventions in an Australian university: a case study. Stress Health. 2015 Feb;31(1):24-34. doi: 10.1002/smi.2517. Epub 2013 Jul 23. PMID 23878071
- [Background] Boscolo P, Di Donato A, Di Giampaolo L, Forcella L, Reale M, Dadorante V, Alparone F, Pagliaro S, Kouri M, Magrini A, Fattorini E. Blood natural killer activity is reduced in men with occupational stress and job insecurity working in a university. Int Arch Occup Environ Health. 2009 May;82(6):787-94. doi: 10.1007/s00420-008-0374-5. Epub 2008 Oct 22. PMID 18941771
- [Background] Neupert SD, Almeida DM, Mroczek DK, Spiro A 3rd. Daily stressors and memory failures in a naturalistic setting: findings from the VA Normative Aging Study. Psychol Aging. 2006 Jun;21(2):424-9. doi: 10.1037/0882-7974.21.2.424. PMID 16768588
- [Background] Aguilar Cordero MJ, Sanchez Lopez AM, Mur Villar N, Garcia Garcia I, Rodriguez Lopez MA, Ortegon Pinero A, Cortes Castell E. [Salivary cortisol as an indicator of physological stress in children and adults; a systematic review]. Nutr Hosp. 2014 May 1;29(5):960-8. doi: 10.3305/nh.2014.29.5.7273. Spanish. PMID 24951973
- [Background] Gao W, Brooks GA, Klonoff DC. Wearable physiological systems and technologies for metabolic monitoring. J Appl Physiol (1985). 2018 Mar 1;124(3):548-556. doi: 10.1152/japplphysiol.00407.2017. Epub 2017 Sep 28. PMID 28970200
- [Background] Mozos OM, Sandulescu V, Andrews S, Ellis D, Bellotto N, Dobrescu R, Ferrandez JM. Stress Detection Using Wearable Physiological and Sociometric Sensors. Int J Neural Syst. 2017 Mar;27(2):1650041. doi: 10.1142/S0129065716500416. Epub 2016 May 16. PMID 27440466
- [Background] Bravo P, Contreras A, Perestelo-Perez L, Perez-Ramos J, Malaga G. [Looking for a more participative healthcare: sharing medical decision making]. Rev Peru Med Exp Salud Publica. 2013 Oct-Dec;30(4):691-7. Spanish. PMID 24448951
- [Background] Peake JM, Kerr G, Sullivan JP. A Critical Review of Consumer Wearables, Mobile Applications, and Equipment for Providing Biofeedback, Monitoring Stress, and Sleep in Physically Active Populations. Front Physiol. 2018 Jun 28;9:743. doi: 10.3389/fphys.2018.00743. eCollection 2018. PMID 30002629
- [Background] Nelson MB, Kaminsky LA, Dickin DC, Montoye AH. Validity of Consumer-Based Physical Activity Monitors for Specific Activity Types. Med Sci Sports Exerc. 2016 Aug;48(8):1619-28. doi: 10.1249/MSS.0000000000000933. PMID 27015387
- [Background] van Hout B, Janssen MF, Feng YS, Kohlmann T, Busschbach J, Golicki D, Lloyd A, Scalone L, Kind P, Pickard AS. Interim scoring for the EQ-5D-5L: mapping the EQ-5D-5L to EQ-5D-3L value sets. Value Health. 2012 Jul-Aug;15(5):708-15. doi: 10.1016/j.jval.2012.02.008. Epub 2012 May 24. PMID 22867780
- [Background] Lee EH. Review of the psychometric evidence of the perceived stress scale. Asian Nurs Res (Korean Soc Nurs Sci). 2012 Dec;6(4):121-7. doi: 10.1016/j.anr.2012.08.004. Epub 2012 Sep 18. PMID 25031113
- [Background] Julian LJ. Measures of anxiety: State-Trait Anxiety Inventory (STAI), Beck Anxiety Inventory (BAI), and Hospital Anxiety and Depression Scale-Anxiety (HADS-A). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S467-72. doi: 10.1002/acr.20561. No abstract available. PMID 22588767
- [Background] Hulley, SB, Cummings SR, Browner WS, Grady DG, Newman TB. Designing Clinical Research. Philadelphia: Lippincott Williams & Wilkins; 2014